CLINICAL TRIAL: NCT06246734
Title: Effect of Companion Robotic Pets on Older Adult Well-Being
Brief Title: Companion Robotic Pets and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Allegheny County Department of Human Services, Area Agency on Aging (Unknown)
Responsible Party: Principal Investigator, Steven M. Albert, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY23090076
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Dementia; Social Behavior; Caregiver Burden
MeSH Terms: conditions — Dementia; Social Behavior; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Single-blind randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor blind to treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment, Immediate Robot Pet Companion (Experimental): Participants will receive a Hasbro Joy for All robotic pet. These are low cost (< $150), life-like cats and dogs that respond to human interaction by making sounds or turning their head for eye contact. The robot companion pets are designed as supports for older people with cognitive impairment. In this trial, the older person can treat it like a pet or ignore it. Family caregivers will report on engagement with the pet and effects on mood.
  Interventions: Behavioral: Hasbro Joy for All robot pet companion
- Control, Delayed Robot Pet Companion (No Intervention): During the 6-8 week trial, this group will not receive the robot pet companion but will complete baseline and follow-up assessments on teh same schedule as the treatment arm. Participants in this arm will receive the robot pet after the trial.

INTERVENTIONS:
Behavioral: Hasbro Joy for All robot pet companion — The robot pets are stuffed animals (dogs and cats) that have features that make them seem lifelike. For example, the animal toys turn their heads when petted, purr or make puppy sounds, feel warm, have a heartbeat, and go to sleep when they are ignored. They respond to attention and petting like a real pet. The robot pets do not collect information and do not require any maintenance, except a battery. Engagement with the device is at the discretion of participants.
  Arms: Treatment, Immediate Robot Pet Companion

SUMMARY:
This research will assess the effect of companion robotic pets on the wellbeing of older adults and their family caregivers.

DETAILED DESCRIPTION:
Social robot pets have been shown to have a positive impact on age-related physical, cognitive, emotional, and social challenges that affect independence and quality of life. These "pets" are designed to interact with people as a real pet might. They purr when stroked, make eye contact, have a heartbeat, turn toward a person when touched, are warm, and appear lifelike. Does introduction of such a pet reduce loneliness or promote engagement in older adults with cognitive or physical disability?

This research will determine if:

1. Older adults with disabilities engage with such robotic companions;
2. Placing a robotic pet in a home enhances mood and positive affect in older people;
3. Caregivers to these adults find the robots beneficial for their own mood and time use.

In a single-blind randomized controlled trial over 6-8 weeks, we hypothesize that older adults in the intervention arm will engage with the pets and show benefit in mood as reported by family caregivers.

ELIGIBILITY:
Inclusion Criteria:

1. Participating in Family Caregiver Support Program or OPTIONS Program administered by Allegheny County Area Agency on Aging
2. Provide unpaid family or friend caregiver support for at least 6 months
3. Older person aged 50+
4. Able to provide verbal informed consent

Exclusion Criteria:

1. Uncomfortable with robot pet companion in home
2. Family Caregiver < 18 years age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2024-03-03 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Positive Affect Scale from Baseline to 6-8 weeks | Baseline and Follow-up, 6-8 weeks later
  PROMIS Positive Affect Short Form 15a Scale: The PROMIS measures are normed for population probability samples, with raw scores transformed into T scores (mean 50, SD=10). The scale measures positive emotion (e.g., enjoyment, engagement, serenity).
Change in Negative Affect from Baseline to 6-8 weeks | Baseline and Follow-up, 6-8 weeks later
  PROMIS Emotional Distress and Anger Short Form Scale: The PROMIS measures are normed for population probability samples, with raw scores transformed into T scores (mean = 50, SD=10). The scale measures emotional distress (e.g., irritability, anger).

OTHER OUTCOMES:
Engagement with Pet | Follow-up interview, 6-8 weeks after baseline
  Adapted companion animal questionnaire, treatment arm. The scale measures daily involvement with a pet, such as the frequency of holding the animal, sleeping in the same room, feeling responsible for the animal). Scale scores range from 6-30.

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Albert, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual-level research data will be made available to qualified researchers who submit an analytic plan for IRB-approved research. Only de-identified data will be shared. Also, we will contact Pitt's Office of Sponsored Programs prior to sharing any data outside of the institution.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Following study completion for 12 months
Access Criteria: Email: smalbert@pitt.edu